CLINICAL TRIAL: NCT02905383
Title: Effect of a Multi-Component Exercise Program on Function and Health in Older People Recently Discharged From Hospital. A Randomized Controlled Clinical Trial.
Brief Title: The Effect of Exercise on Physical Function and Health in Older People After Discharge From Hospital
Acronym: OLPADIS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oslo Metropolitan University (Other)
Responsible Party: Principal Investigator, Sylvia Sunde, Phd-student, Oslo Metropolitan University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 2015/2432
Record Dates: First submitted 2016-09-05; First posted 2016-09-19 (Estimated); Last update posted 2020-08-04 (Actual); Status verified 2020-08

CONDITIONS: Chest Pain; Pneumonia; Transient Ischemic Attack; Stroke; Functional Failure
MeSH Terms: conditions — Chest Pain; Pneumonia; Ischemic Attack, Transient; Stroke | interventions — Exercise

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Exercise (Experimental): This group will perform a multi-component exercise program twice a week for 16 weeks. The multi-component exercise program consists of endurance training, progressive strength exercises and balance exercises. The intervention will be individualised, but performed in groups of four to ten patients. The participants are also expected to do exercises on their own, at least once weekly.
  Interventions: Other: Exercise
- Control (No Intervention): The participants in the control group will be encouraged to exercise on their own, according to the World Health Organization recommendations on physical activity for adults aged 65 and above.

INTERVENTIONS:
Other: Exercise — A multi-component exercise program that consists of endurance training, progressive strength exercises and balance exercises.
  Arms: Exercise

SUMMARY:
The aim of this study is to investigate the effect of a multi-component exercise program on physical function, physical activity and health-related quality of life (HRQOL) in older people recently discharged from hospital. The intervention consists of 32 group-based exercise sessions, performed twice a week. In addition the participants in the intervention group will be encouraged to perform an exercise program on their own, at least once weekly. The participants in the control group will be encouraged to exercise on their own, according to the World Health Organization (WHO) recommendations on physical activity for adults aged 65 and above.

DETAILED DESCRIPTION:
Older people who have been hospitalized often experience loss of function, increased risk of falls and reduced health-related quality of life (HRQOL) in the post-discharge period. The reason for this is the cumulative effect of illness, bedrest during hospital stay and inactivity after discharge. Previous research indicates that exercise therapy should be an integrated part of the post-hospital treatment to prevent or postpone this functional decline and improve HRQOL. Therefore, the investigators will conduct a randomized controlled trial to investigate the effect of a multi-component exercise program consisting of high intensity exercises on physical function, physical activity and HRQOL among older people living at home after discharge from hospital after treatment of an acute medical event.

ELIGIBILITY:
Inclusion Criteria:

* 65 years or older, live in their own home, consent to participate in the program three times a week (twice a week outside their home), manage to walk with or without assistive device, and assessed by a doctor as able to tolerate the intervention.

Exclusion Criteria:

* Severe cognitive impairment (Mini-Mental State Examination (MMSE) score less than 20), have an expected lifespan less than one year, exercise more than twice a week, and score above nine points on the Short Physical Performance Battery.

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 88 (Actual)
Dates: Start 2016-09-29; Primary Completion 2020-01-30 (Actual); Study Completion 2020-01-30 (Actual)

PRIMARY OUTCOMES:
Changes in physical function | Baseline, 4 months and 8 months
  Changes in physical function will be measured with The Short Physical Performance Battery (SPPB). This test evaluates balance, mobility and muscle strength by examining an individual's ability to stand with feet together side-by side, semitandem and tandem positions, time to walk 8ft and time to rise from a chair and return to the seated position five times. Each of the three tests is scored, based on performance between 0 and 4, leaving a maximum score of 12 for those individuals performing at the highest levels.

SECONDARY OUTCOMES:
Berg Balance Scale | Baseline, 4 months and 8 months
  Berg Balance Scale is a measure of performance-based balance. It comprises 14 observable tasks frequently encountered in everyday life.
Health-related quality of life (HRQOL) | Baseline, 4 months and 8 months
  HRQOL measured by the Medical Outcome Study 36 Item Short-Form Health Survey (SF-36)
Physical Activity measured by the short form of the International Physical Activity Questionnaire (IPAQ-SF) | Baseline, 4 months and 8 months
  The IPAQ-SF includes seven questions about the time spent in vigorous- and moderate intensity activities, walking and sedentary activity.
Muscle mass | Baseline, 4 months and 8 months
  Muscle mass will be measured by bioimpedance
Compliance to the intervention | Eight months from baseline
  Participants will complete an activity diary where they are asked to report completion of exercise, non-protocol activity and any adverse events related to the exercise. Patients are considered non-compliant if they have undertaken less than 50% of the prescribed exercise.
Feasibility of the intervention | Four months from baseline
  Adverse events will be registered as outlined by Oryet al. (2005) in the following four categories: falls, cardiovascular events, musculoskeletal injuries and health care utilization.
Amount of home-help services received | Baseline, 4 months and 8 months
  If they receive any home care
Handgrip strength | Baseline, 4 months and 8 months
  Handgrip strength in kilograms measured using a hydraulic dynamometer
Height | Baseline
  Height will be measured in meters

CONTACTS AND LOCATIONS:
Overall Officials: Therese Brovold, Phd, Principal Investigator — Oslo University College of Applied Science
Locations (1):
- Diakonhjemmet Hospital, Oslo, Norway

REFERENCES:
- [Derived] Sunde S, Hesseberg K, Skelton DA, Ranhoff AH, Pripp AH, Aaronaes M, Brovold T. Associations between health-related quality of life and physical function in older adults with or at risk of mobility disability after discharge from the hospital. Eur Geriatr Med. 2021 Dec;12(6):1247-1256. doi: 10.1007/s41999-021-00525-0. Epub 2021 Jun 9. PMID 34106446
- [Derived] Sunde S, Hesseberg K, Skelton DA, Ranhoff AH, Pripp AH, Aaronaes M, Brovold T. Effects of a multicomponent high intensity exercise program on physical function and health-related quality of life in older adults with or at risk of mobility disability after discharge from hospital: a randomised controlled trial. BMC Geriatr. 2020 Nov 11;20(1):464. doi: 10.1186/s12877-020-01829-9. PMID 33176703